CLINICAL TRIAL: NCT05598242
Title: Amniotic Membrane Treatment for Hyposecretory Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Principal Investigator, Emiliano Facundo Ross, Medical doctor, Hospital Nacional Profesor Alejandro Posadas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192 LUPeSe/18 (ENM)
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Dry Eye Syndromes; Sjogren Syndrome With Keratoconjunctivitis
Keywords: dry eye; autologous serum; amniotic membrane extract eye drops
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: active-controlled, parallel-group trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane extract (Experimental): patients receive amniotic membrane eye drops (AMEED) as 1 drop in each eye 6 times daily, 30 days
  Interventions: Biological: Amniotic membrane extract eye drops (AMEED)
- autologous serum eye drops (Active Comparator): patients receive autologous serum eye drops (ASED) as 1 drop in each eye 6 times daily, 30 days
  Interventions: Biological: Amniotic membrane extract eye drops (AMEED)

INTERVENTIONS:
Biological: Amniotic membrane extract eye drops (AMEED) — Following a 2-week wash out period, patients were allocated randomly to receive AMEED, administered as 1 drop in each eye 6 times daily, respectively, for 30 days.
  Other Names: Autologous serum

SUMMARY:
The goal of this randomized, active-controlled, parallel-group trial is to evaluate the clinical efficacy of amniotic membrane extract eye drops (AMEED) in reducing signs and symptoms of hyposecretory dry eye

Participants will receibed amniotic membrane extract eye drops 6 times daily and was evaluated at baseline day and day 30th.

Researchers will compare against autologous serum eye drops effects

DETAILED DESCRIPTION:
This was a randomized, active-controlled, parallel-group trial. The perfect masked conditions could not be accomplished because the autologous serum eye drops needs venous punction for it preparation.

During de initial 2 weeks screening period, the patients received artificial tears 4 times daily to minimize the effects of any eye drops used before patients were allocated randomly to receive autologous serum eye drops (ASED) or AMEED, administered as 1 drop in each eye 6 times daily, respectively, for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* dry eye related symptoms
* Fluorescein Corneal Staining score of 4 or more
* Lisamina Green Conjunctival score of 4 or more
* a no-anesthesia Schirmer test value at 5' of 10 mm or less

Exclusion Criteria:

* glaucoma treatment
* surgical procedures within 3 months of the baseline evaluation
* precense of punctal plug
* patients that were human immunodeficiency virus positive

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — frecuency of the illness
Enrollment: 37 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Lisamina green conjunctival staining | 1 month
  changes in the lisamina green conjunctival staining (LGCS) score to demonstrate ocular surface damage

SECONDARY OUTCOMES:
Fluorescein Corneal staining | 1 month
  fluorescein corneal staining (FCS) score to demostrate corneal ephithelium involment
Schirmer's test | 1 month
  Schirmer´s test to asses lacrimal production whithout anesthesia
TBUT | 1 month
  tear film break up time
OSDI | 1 month
  severity of symptoms reported by patients according to the ocular surface disease index (OSDI)

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano F Ross, MD, Principal Investigator — assistant
Locations (3):
- Argentina (3):
  - Hospital Nacional Posadas, El Palomar, Buenos Aires
  - Hospital Nacional Prof. A. Posadas, El Palomar, Buenos Aires
  - Hospital Nacional Profesor A. Posadas, El Palomar, Buenos Aires

IPD SHARING:
Plan to Share IPD: No